CLINICAL TRIAL: NCT01632085
Title: Comparison of Two Laryngoscopes: Single-use Device Laryngobloc ® (SU) Versus Reusable Handle With Disposable Metal Blade (R) : Quality of Laryngoscopy and Bacterial Contamination of the Handle
Brief Title: Comparison of Two Laryngoscopes: Single-use Device Laryngobloc ® (SU) Versus Reusable Handle With Disposable Metal Blade (R)
Acronym: MUUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5131; 2011-A01548-33 (Other: ANSM)
Record Dates: First submitted 2012-06-21; First posted 2012-06-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Contamination of the Handles; Quality of the Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group SU (Single use or Laryngobloc ®) ®) (Other): In order to avoid an order effect, the patient acting as his own control, will randomly undergo a laryngoscopy with each laryngoscopes, the intubation being performed during the second laryngoscopy, here with the Laryngobloc ®.
  Interventions: Device: The two groups SU and R are defined by the device with which intubation is performed after a first laryngoscopy done with the other device.
- Group R (Reusable handle) (Other): In order to avoid an order effect, the patient acting as his own control, will randomly undergo a laryngoscopy with each laryngoscopes, the intubation being performed during the second laryngoscopy, here with the Disposable Metal Blade.
  Interventions: Device: The two groups SU and R are defined by the device with which intubation is performed after a first laryngoscopy done with the other device.

INTERVENTIONS:
Device: The two groups SU and R are defined by the device with which intubation is performed after a first laryngoscopy done with the other device. — Group SU (Single Use or Laryngobloc ®): the first laryngoscopy is performed with the R and the second laryngoscopy and the intubation is performed with the Laryngobloc ®.
  Group R (Reusable handle+ disposable metal blade): the first laryngoscopy is performed with the Laryngobloc ® and the second laryngoscopy and the intubation is performed with the R.

SUMMARY:
Reduce the risk of nosocomial transmission of germs related to the reusability of the laryngoscope handle. The alternative is to replace it with a disposable device, provided that it is as effective as the reference strategy at a reasonable cost.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years·
* Hospitalized for elective surgery and targeted for orotracheal intubation under direct laryngoscopy under general anesthesia with neuromuscular blockade resolved·
* Subject has signed informed consent·
* Suject affiliated to a social protection·
* Subject informed of the results of medical examination

Exclusion Criteria:

* Contraindication to general anesthesia or one of its components·
* General anesthesia without a competitive muscle relaxant·
* Patient with criteria for difficult intubation·
* Patient targeted for special care of the airway (fiberoptic or vidéolaryngoscopy), whatever the indication as Mallampati class 4·
* Subject in class 4 Mallampati·
* Acts performed in the emergency setting·
* Pregnancy and obstetric procedures·
* Breastfeeding·
* Difficulty in communication with the patient (including obtaining informed consent, evaluation of pain in the recovery Room ·
* Subject in exclusion period (determined by a previous study or a study in progress)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The quality of laryngoscopy | 1 year
  The quality of laryngoscopy. The quality of the visibility of the glottis, is assessed by the Cormack and Lehane grade. A rank of 1 or 2 will be considered a success for the analysis of results.

SECONDARY OUTCOMES:
Evaluation microbiological and evaluation of intubation | 1 year
  Evaluation microbiological (bacteria, fungi) and identification of bacteria with smears of the handle of laryngoscopes, the Laryngobloc ® and the reusable battery.
  Evaluation of intubation: IDS score, satisfaction of the anesthesiologist, intubation time, quality of light offered by the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France